CLINICAL TRIAL: NCT05072873
Title: The Adjunctive Role of Temporary Uterine Packing Combined With Topical Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Women With Twin Pregnancy Undergoing Cesarean Section: A Randomized Controlled Trial
Brief Title: Topical Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Women With Twin Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/543/7/21
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: a double-blind randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blind randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical tranexamic acid (Experimental): temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid
  Interventions: Drug: Topical tranexamic acid
- normal saline (Placebo Comparator): temporary uterine packing with gauze of the dimensions soaked with 2 gm placebo to tranexamic diluted in 60ml saline acid
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Topical tranexamic acid — temporary uterine packing with gauze of the dimensions soaked with 2 gm tranexamic diluted in 60ml saline acid
  Other Names: experimental
  Arms: Topical tranexamic acid
Other: normal saline — temporary uterine packing with gauze of the dimensions soaked with 2 gm placebo to tranexamic diluted in 60ml saline acid
  Other Names: Placebo Comparator
  Arms: normal saline

SUMMARY:
twin pregnant women requesting cesarean section, the effectiveness and safety of temporary uterine packing coupled with topical tranexamic acid as an adjuvant for decreasing blood loss during delivery were compared to placebo.

DETAILED DESCRIPTION:
The most common cause of postpartum hemorrhage (PPH) is uterine atony, which accounts for up to 80% of PPH occurrences. PPH is the main cause of maternal morbidity and mortality, accounting for up to 28% of all maternal deaths globally. As a result, generating a fast and efficient uterine contraction after birth is critical. Obesity, White or Hispanic race/ethnicity, polyhydramnios, preeclampsia, anemia, and chorioamnionitis, as well as a twin pregnancy, are all risk factors for uterine atony.

ELIGIBILITY:
Inclusion Criteria:

* Women With Twin Pregnancy Undergoing Cesarean Section

Exclusion Criteria:

* Patients with cardiac, hepatic, renal, or thromboembolic disease. ,
* patients with a high possibility of the morbid adherent placenta,
* known coagulopathy and
* those presented with severe antepartum hemorrhage
* refuse to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women With Twin Pregnancy Undergoing Cesarean Section
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | 30 minutes
  measurement the intraoperative blood loss by direct and gravimetric methods

SECONDARY OUTCOMES:
postoperative blood loss | 12 hours
  measurement the intraoperative blood loss by direct and gravimetric methods
need of blood transfusion | 24 hours
  number of unites of blood transfusion
need of uterotonic | 24 hours
  misoprostol, oxytocin etc
change in hemoglobin | 24 hours
  change in hemoglobin

IPD SHARING:
Plan to Share IPD: No